CLINICAL TRIAL: NCT01719666
Title: Randomized Control Trial on Lateral Retinaculum Release in MPFL Reconstruction
Brief Title: Medial Patellofemoral Ligament Reconstruction With or Without Lateral Retinaculum Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010.651
Record Dates: First submitted 2011-12-22; First posted 2012-11-01 (Estimated); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Episodic Patellar Dislocation
Keywords: MPFL; patella; dislocation; release
MeSH Terms: conditions — Patella Fracture; Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- isolated MPFL reconstruction (Other)
  Interventions: Procedure: conventional surgery
- MPFL reconstruction and Lateral retinaculum release (Experimental)
  Interventions: Procedure: MPFL reconstruction and lateral retinaculum release

INTERVENTIONS:
Procedure: MPFL reconstruction and lateral retinaculum release — MPFL is performed with a standard technique using gracilis tendon. A tunnel is performed at the femoral part with a bioabsorbable screw fixation and 2 bundles with suture fixation at the patellar side
  Arms: MPFL reconstruction and Lateral retinaculum release
Procedure: conventional surgery — conventional surgery: MPFL reconstruction
  Arms: isolated MPFL reconstruction

SUMMARY:
The investigators hypothesis is lateral retinaculum release has no effect on treatment of Patellar Recurrent Dislocation with Medial Patellofemoral Ligament (MPFL) reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* age between 18yo and 45yo
* indication for MPFL reconstruction
* unilateral or bilateral indication

Exclusion Criteria:

* indication for bony procedures
* previous surgery for PF disorders
* patient refusal

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2011-11-22 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Patellar tilt measurement | 2 years of follow up
  IKDC score, patellar tilt measurement on x-rays and CT-scan

SECONDARY OUTCOMES:
rate of complications | 2 years of follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Faure F, Erard J, Batailler C, Magnussen RA, Lustig S, Servien E. Lateral Retinacular Release During MPFL Reconstruction: A Randomized Clinical Trial. Am J Sports Med. 2025 Oct;53(12):2869-2874. doi: 10.1177/03635465251366306. Epub 2025 Sep 11. PMID 40934533